CLINICAL TRIAL: NCT01981447
Title: IV Lacosamide: The Safety of Intravenous Lacosamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, James W. Wheless, Principal Investigaor, Neurolgy Division Chief, Le Bonheur Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-00570-FB
Record Dates: First submitted 2013-05-13; First posted 2013-11-11 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): IV Lacosamide administered (intravenously) over 30 minutes: 0.7mg/kg, 1.4 mg/kg, 2.1 mg/ kg and 2.9 mg/kg over 30 minutes.
  Interventions: Drug: IV Lacosamide
- Group B (Active Comparator): IV Lacosamide to be administered (intravenously) over 15 minutes: 0.7mg/kg, 1.4 mg/kg, 2.1mg/kg, 2,4 mg/kg
  Interventions: Drug: IV Lacosamide

INTERVENTIONS:
Drug: IV Lacosamide — Lacosamide administered intravenously over 15 or 30 minutes, depending on study arm, to patients with epilepsy.
  Other Names: Vimpat

SUMMARY:
The purpose of this study is to evaluate the safety of IV Lacosamide in children ages 4-35.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety of IV Lacosamide in children ages 4 years to 35 years, inclusive who are unable to take oral medications or require parenteral administration of IV Lacosamide Occasionally, patients over the age of 20 are seen at LeBonheur Children's Hospital due to the complexity of their condition, or due to a long relationship with their physician. These are exceptions which are reviewed on a case by case basis and are approved by the hospital administrator for admissions and outpatient testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient or LAR must sign informed consent
* Diagnosis of partial onset currently uncontrolled
* Patient must have received anti-epileptic drug therapy prior to initiation
* Patient must have a medical condition in which parental administration is desireable
* Male or female
* Ages 4-35

Exclusion Criteria:

* Patient has participated in a study involving IV Lacosamide
* Patient has had an episode of status epilepticus in the last 3 months
* Drug history to lacosamide pregnant or lactating
* If of child bearing age, must have pregnancy test
* Patient has participated in an experimental drug study in last 30 days
* Patients with significant active hepatic or renal disease.
* Patients with known cardiac disease.

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (TEAEs), reported or observed. | 2 years
  Bradycardia, hypotension, fatigue, nausea, somnolence.
Measure post-infusion lacosamide plasma concentrations | 2 years
  Serum lacosamide level drawn from the arm opposite intravenous infusion
Measure changes in EKG, PR interval | 2 years
  PR interval changes measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: James W Wheless, MD, Principal Investigator — Lebonheur Children's Medical Center
Locations (1):
- Lebonheur Children's Hospital, Memphis, Tennessee, United States